CLINICAL TRIAL: NCT02189434
Title: A Pilot Study to Determine the Correlation of Serum Procalcitonin Levels and Development of Sepsis in Patients Undergoing Cytoreductive Surgery
Brief Title: Does Serum Procalcitonin Levels Predict Sepsis in Patients Undergoing Cytoreductive Surgery
Status: Completed | Type: Observational
Sponsor: Eastern Regional Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: ERMC 14-14
Record Dates: First submitted 2014-07-10; First posted 2014-07-14 (Estimated); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: Cytoreductive Surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Collection of serum blood specimens
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cytoreductive surgery: Patients having undergone cytoreductive surgery with or without HIPEC will have serum procalcitonin lab draws
  Interventions: Other: Serum procalcitonin lab draws

INTERVENTIONS:
Other: Serum procalcitonin lab draws — Blood will be collected in a 4mL capacity, green top lithium heparin tube. Samples can be drawn from a port with other labs. The samples will be centrifuged and then the plasma/serum will be removed and placed into a screw-capped round bottom plastic vial. Samples will be stored at -20○C until processing. Serum samples will be batch processed for each participant at the conclusion of their study period.
  These draws will be conducted for the sole purpose of this study, and whenever possible, they will be performed at the same time as routine blood draws conducted for medical monitoring to reduce the burden to the patients.

SUMMARY:
Serum procalcitonin levels will be considerably higher, for a longer period of time, in patients who develop sepsis compared to patients with SIRS or those who have an uncomplicated post-surgical recovery. Monitoring of serum procalcitonin trends will allow for an earlier diagnosis of, and initiation of treatment for, sepsis compared to current standard ICU methods.

ELIGIBILITY:
Inclusion Criteria:

* Female or male person ≥ 18 years of age
* Biopsy proven carcinoma
* Scheduled for cytoreductive surgery, with or without HIPEC
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) = 0, 1, or 2
* Able to give informed consent for protocol participation

Exclusion Criteria:

* Participants are not able to understand or provide written informed consent
* Pre-operative anti-inflammatory medication use within 72 hours of their baseline blood draw
* Pre-operative infection treatment with corticosteroids within 72 hours of their baseline blood draw
* Immunosuppressive illness other than neoplasm
* Pregnant or lactating female

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients having undergone cytoreductive surgery with or without HIPEC
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-06; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to determine the natural progression of serum procalcitonin in patients recovering from cytoreductive surgery, with or without HIPEC. | end of study

SECONDARY OUTCOMES:
Observe the patient's post-operative course with regards to serum procalcitonin levels and development of sepsis in patients previously treated with cytoreductive surgery with or without HIPEC. | end of study

CONTACTS AND LOCATIONS:
Overall Officials: Rod Flynn, MD, Principal Investigator — Eastern Regional Medical Center
Locations (1):
- Eastern Regional Medical Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided